CLINICAL TRIAL: NCT04561518
Title: ConTTRibute: A Global Observational Multicenter Long-Term Study of Patients With Transthyretin (TTR)-Mediated Amyloidosis (ATTR Amyloidosis)
Brief Title: ConTTRibute: A Global Observational Study of Patients With Transthyretin (TTR)-Mediated Amyloidosis (ATTR Amyloidosis)
Acronym: ConTTRibute
Status: Recruiting | Type: Observational
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-TTR02-013
Record Dates: First submitted 2020-09-18; First posted 2020-09-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Transthyretin-Mediated Amyloidosis; ATTR Amyloidosis
Keywords: RNAi therapeutic; Transthyretin; TTR; Amyloidosis; Hereditary Transthyretin-mediated (hATTR) Amyloidosis; hATTR amyloidosis; Hereditary ATTR amyloidosis; Wild-type amyloidosis; wtATTR amyloidosis; ATTRv amyloidosis; ATTRwt amyloidosis; Polyneuropathy; Familial amyloid polyneuropathies; ATTR; Transthyretin amyloidosis; TTR-mediated amyloidosis; Polyneuropathies; Amyloid neuropathies; Amyloid neuropathies, familial; Amyloidosis, familial
MeSH Terms: conditions — Amyloidosis; Amyloid Neuropathies, Familial; Polyneuropathies; Amyloidosis, Hereditary, Transthyretin-Related; Amyloid Neuropathies; Amyloidosis, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ATTR amyloidosis: Patients with a diagnosis of ATTR amyloidosis, hereditary or wild type, will be eligible for the study and will follow routine clinical care.
- Pre-symptomatic Carriers: Pre-symptomatic carriers with a known disease-causing TTR variant will be eligible for the study and will follow routine clinical care.

SUMMARY:
The purpose of this study is to:

* Describe epidemiological and clinical characteristics, natural history and real-world clinical management of ATTR amyloidosis patients
* Characterize the safety and effectiveness of patisiran and vutrisiran as part of routine clinical practice in the real-world clinical setting
* Describe disease emergence/progression in pre-symptomatic carriers of a known disease-causing transthyretin (TTR) variant

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ATTR amyloidosis or documented known disease-causing TTR variant for the cohort of pre-symptomatic carriers
* Germany Only: Patients must be treated per the summary of product characteristics (SmPC) for any approved treatment for ATTR amyloidosis

Exclusion Criteria:

* Current enrollment in a clinical trial for any investigational agent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of ATTR amyloidosis, hereditary or wild type, and pre-symptomatic carriers with a known disease-causing TTR variant will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | From time of enrollment for up to 10 years
Selected Events of Interest in Patients with Hereditary Transthyretin-mediated (hATTR) Amyloidosis (ATTRv Amyloidosis) | From 1 year prior to enrollment for up to 10 years
  Selected events of interest are defined as hepatic events, cardiovascular events, renal events, ocular events and infusion-related reactions, hypersensitivity, and other events in patients diagnosed with hATTR amyloidosis.
Health Care Provider (HCP)-Assessed Polyneuropathy (PND) Disability Score | Up to 11 years
  PND Scores: Stage 0=No symptoms; Stage I=Sensory disturbances but preserved walking capabilities; Stage II=Impaired walking capacity, but ability to walk without a stick or crutches; Stage IIIA=Walking with help of 1 stick or crutch; Stage IIIB=Walking with the help of 2 sticks or crutches; Stage IV=confined to wheel chair or bedridden.
HCP-Assessed Familial Amyloidotic Polyneuropathy (FAP) Score | Up to 11 years
  FAP Scores: Stage 0=No symptoms; Stage I=Unimpaired ambulation; mostly mild sensory, motor and autonomic neuropathy in the lower limbs; Stage II=Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk; Stage III=Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs.
HCP-Assessed Neuropathy Impairment Score (NIS) | Up to 11 years
  NIS : 74 items, assess muscle weakness, reflexes and sensation; scored separately for left, right limbs (37 items for each side). Components of muscle weakness (hip and knee flexion, hip and knee extension, ankle dorsiflexors, ankle plantar flexors, toe extensors, toe flexors) scored on scale 0 (normal) to 4 (paralysis), higher score=greater weakness. Components of reflexes (quadriceps femoris, triceps surae) and sensation (touch pressure, pin-prick, vibration, joint position) scored 0 = normal, 1= decreased, or 2 = absent. Total possible NIS score range 0-244, higher score=greater impairment.
HCP-Assessed Cardiomyopathy | Up to 11 years
  Cardiomyopathy will be assessed using New York Heart Association (NYHA) Class: I=No symptoms; II=Symptoms with ordinary physical activity; III=Symptoms with less than ordinary physical activity; IV=Symptoms at rest.
HCP- Assessed Cardiopulmonary Exercise Testing (CPET) Performance | Up to 11 years
Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) Total Score | Up to 11 years
  Norfolk-QoL-DN: The Norfolk QOL-DN questionnaire is a standardized 35-item patient-reported outcomes measure that assesses 6 domains: physical function, large-fiber neuropathy, activities of daily living, symptoms, small-fiber neuropathy, and autonomic neuropathy. The total score ranges from -4 points (best possible quality of life) to 136 points (worst possible quality of life).
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Up to 11 years
  The KCCQ is a 23-item self-administered questionnaire developed to independently measure the patient's perception of health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life within a 2-week recall period. The KCCQ quantifies 6 domains (symptoms, physical function, quality of life, social limitation, self-efficacy, and symptom stability) and 2 summary scores (clinical and overall summary [OS] scores).
Rasch-built Overall Disability Scale (R-ODS) | Up to 11 years
  The R-ODS is a 24-item self-administered questionnaire for assessment of the disability a patient experiences. It uses a linearly weighted categorical rating scale that specifically captures domains of activity and social participation limitations in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (40):
- United States (13):
  - Clinical Trial Site, La Jolla, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Iowa City, Iowa
  - Clinical Trial Site, Kansas City, Kansas
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Austin, Texas
  - Clinical Trial Site, Houston, Texas
- Brazil (2):
  - Clinical Trial Site, Salvador
  - Clinical Trial Site, São Paulo
- Clinical Trial Site, Sofia, Bulgaria
- Denmark (2):
  - Clinical Trial Site, Aarhus
  - Clinical Trial Site, Copenhagen
- France (5):
  - Clinical Trial Site, Bordeaux
  - Clinical Trial Site, Bron
  - Clinical Trial Site, Créteil
  - Clinical Trial Site, Le Kremlin-Bicêtre
  - Clinical Trial Site, Marseille
- Germany (3):
  - Clinical Trial Site, Berlin
  - Clinical Trial Site, Giessen
  - Clinical Trial Site, Hanover
- Israel (2):
  - Clinical Trial Site, Jerusalem
  - Clinical Trial Site, Ramat Gan
- Italy (4):
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Naples
  - Clinical Trial Site, Palermo
  - Clinical Trial Site, Roma
- Clinical Trial Site, Groningen, Netherlands
- Portugal (2):
  - Clinical Trial Site, Lisbon
  - Clinical Trial Site, Porto
- Spain (3):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Palma
- Taiwan (2):
  - Clinical Trial Site, New Taipei City
  - Clinical Trial Site, Taipei

IPD SHARING:
Plan to Share IPD: No